CLINICAL TRIAL: NCT04504669
Title: A Phase I First-in-Human Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of AZD8701 Administered Intravenously as Monotherapy and in Combination With Durvaluamb (MEDI4736) in Participants With Advanced Solid Tumours.
Brief Title: First Time in Human Study of AZD8701 With or Without Durvalumab in Participants With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9950C00001; 04504669 (Other: NCT number); 2019-004539-22 (EudraCT Number)
Record Dates: First submitted 2020-07-16; First posted 2020-08-07 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Clear Cell Renal Cell Cancer; Non-Small-Cell Lung Cancer; Triple Negative Breast Neoplasms; Squamous Cell Cancer of Head and Neck; Small Cell Lung Cancer; Gastroesophageal Cancer; Melanoma; Cervical Cancer; Advanced Solid Tumours
Keywords: Solid Tumours; Durvalumab; MEDI4736; AZD8701; Non Small cell Lung cancer; ccRenal Cancer; TNBC; first time in human; PD-L1; T regulatory cells; FOXP3
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Small Cell Lung Carcinoma; Melanoma; Uterine Cervical Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: This is a Phase I, FIH, multicentre, open-label, multiple arm study. Dose-escalation will occur with AZD8701 in monotherapy and in combination with durvalumab in selected participants with HNSCC, TNBC, NSCLC, ccRCC, gastroesophgeal cancer, melanoma, cervical cancer, small-cell lung cancer and/or participants with solid tumours who have demonstrated a response to prior PD-(L)1 treatment.
  Disease specific expansions will occur with a selected dose of AZD8701 in participants with NSCLC and with a selected dose of AZD8701 and durvalumab in participants with TNBC and clear cell RCC.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): Participants will receive AZD8701 intravenously, on Day 1, 3, 5 and 8 and then weekly for a maximum of 2 years.
  Interventions: Drug: AZD8701
- Combination Therapy (Experimental): Participants will receive AZD8701 (intravenously, on Day 1, 3, 5 and 8 and then weekly) and durvalumab (MEDI4736) intravenously monthly for a maximum of 2 years.
  Interventions: Drug: AZD8701; Biological: Durvalumab

INTERVENTIONS:
Drug: AZD8701 — FOXP3 antisense oligonucleotide
Biological: Durvalumab — anti PDL-1 monoclonal antibody
  Other Names: MEDI4736
  Arms: Combination Therapy

SUMMARY:
The purpose of this study is to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Antitumor Activity of AZD8701 Alone and in Combination with Durvalumab (MEDI4736) in Adult Subjects with Select Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a Phase I, First in Human, multicentre, open-label, multiple arm study with dose escalations and expansions at selected doses. Dose-escalation will occur with AZD8701 in monotherapy (Part 1) and in combination with durvalumab (Part 3) in selected participants with HNSCC, TNBC, NSCLC, ccRCC, gastroesophageal cancer, melanoma, cervical cancer, small-cell lung cancer and/or participants with solid tumours who have demonstrated a response to prior PD-(L)1 treatment.

Disease specific expansions will occur with a selected dose of AZD8701 in participants with NSCLC (Part 2) and with a selected dose of AZD8701 and durvalumab in participants with TNBC and clear cell RCC (Part 4).

ELIGIBILITY:
Inclusion Criteria:

The study is comprised of 2 main parts Monotherapy (AZD8701) and Combined Therapy (AZD8701 and Durvalumab).

Inclusion criteria Dose escalation stages:

* Histological or cytological confirmation of a solid, malignant tumour including HNSCC, TNBC, NSCLC, ccRCC, gastroesophageal cancer, melanoma, cervical cancer, SCLC, and/or participants with other solid tumours who have demonstrated a response to prior anti-PD-(L)1 treatment
* Participant with progressive disease that is refractory to standard therapies or for which no standard therapies exist and a clinical trial is the best option for next treatment based on prior response and/or tolerability to standard of care

Inclusion Criteria Dose Expansions:

Non Small Lung Cancer Participants who have received prior PD(L)1 treatment. Clear Cell Renal Cancer Participants who have not received prior PD(L)1 treatment.

Triple negative Breast Cancer participants who have who have not received prior PD(L)1 treatment.

General inclusion criteria:

* Must be 18 year old at the time of screening
* Body weight > 35 kg
* Male and Female participants of childbearing potential must use effective methods of contraception
* Capable of giving signed informed consent
* ECOG performance status of 0 to 1
* A serum albumin > 30g/L
* Life expectancy of > 12 weeks
* At least 1 lesion, that qualifies as a RECIST 1.1 target lesion at baseline. Tumour assessment by CT scan or MRI must be performed within 28 days prior to treatment.
* Participants must provide a new or previous tumour sample
* Adequate organ system functions

Exclusion Criteria:

* A condition that, in the opinion of the Investigator, would interfere with evaluation of the study intervention or interpretation of participant safety or study results
* History of allogeneic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders Uncontrolled intercurrent illness
* Significant cardiac disease
* History of another primary malignancy except for

  1. Malignancy treated with curative intent and with no known active disease ≥ 5 years
  2. non-melanoma skin cancer
  3. Adequately treated carcinoma in situ without evidence of disease.
* Participant with previous or confirmed Covid 19 diagnosis requiring significant medical intervention
* Current clinical signs and symptoms consistent with COVID-19 or confirmed current infection by appropriate laboratory test within the last 4 weeks prior to screening
* Any major unresolved toxicity from previous anticancer therapy
* Known allergy or hypersensitivity to any of the study interventions or any of the study intervention excipients.

Prior/Concomitant Therapy

* Receipt of the last dose of anticancer therapy within 5 half-lives or ≤ 21 days prior to the first dose of study
* Prior treatment with potential Treg depletion therapies including agents targeting OX40 or CD357 (GITR) for 90 days prior to enrolment on study.
* Participants who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4:

  1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
  2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline
  3. Must not have experienced a ≥ Grade 3 imAE or a neurologic or ocular imAE of any grade while receiving prior immunotherapy.
  4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug. b. The following are exceptions to this criterion:

  1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection).
  2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment
* Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study intervention.
* Major surgical procedure within 28 days prior to the first dose
* Participants receiving anticoagulation therapy with vitamin K antagonists (eg warfarin)
* Participation in another clinical study with study intervention administered in the last 30 days
* Female participants who are pregnant or breastfeeding or male and female participants of reproductive potential who are not willing to employ effective birth control

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated dose (or optimal dose or maximum feasible dose) and RP2D of AZD8701 as monotherapy and in combination with Durvalumab assessed through evaluation of AEs and SAEs | From screening until 105 days after last dose of study treatment
  Determined according to Incidence and treatment related AEs and SAEs
Maximum Tolerated dose (or optimal dose or maximum feasible dose) and RP2D of AZD8701 as monotherapy and in combination with Durvalumab assessed through evaluation of Dose Limiting Toxicities (DLTs) | First 28 day cycle
  Determined according to Incidence of DLTs (during the first 28 day cycle)
Maximum Tolerated dose (or optimal dose or maximum feasible dose) and RP2D of AZD8701 as monotherapy and in combination with Durvalumab assessed through evaluation of vital signs and abnormal laboratory parameters | From screening until 105 days after last dose of study treatment
  Determined according to Incidence of abnormal vital signs and laboratory parameters
Incidence of AEs and SAEs related to AZD8701 as monotherapy and in combination with Durvalumab in disease specific expansions treated at the MTD/OBD/MFD | From screening until 105 days after last dose of study treatment
  Safety and tolerability of the MTD/OBD/MFD assessed through incidence of AEs and SAEs
Objective Response Rate according to RECIST 1.1 by investigator assessment in disease specific expansions treated at the MTD/OB/MFD | Every 8 weeks (first 48 weeks) and then every 12 weeks from start of treatment until the earlier of progression, death, start of subsequent anti-cancer therapy or end of study (for max 42 months)
  The proportion of subjects achieving a confirmed complete or partial response according to RECIST 1.1 by investigator assessment

SECONDARY OUTCOMES:
Progression-free survival according to RECIST 1.1 by investigator assessment | every 8 weeks (first 48 weeks) and then every 12 weeks from start of treatment until the earlier of progression, death or end of study (for max 42 months)
  Time from start of study treatment to the date of objective disease progression or death (by any cause in the absence of progression)
Duration of Response according to RECIST 1.1 by investigator assessment | every 8 weeks (first 48 weeks) and then every 12 weeks from start of treatment until the earlier of progression, death or end of study (for max 42 months)
  Time from first documented response (that is subsequently confirmed) to the date of objective disease progression or death (by any cause in the absence of progression)
Disease Control Rate at 16 weeks according to RECIST 1.1 by investigator assessment | Every 8 weeks from start of treatment until earlier of progression, death or start of subsequent anti-cancer therapy (for up to 24 weeks). Subjects followed to 24 weeks for assessment of SD for 16 weeks from first tumour assessment at 8 weeks
  The proportion of subjects with a best response of CR or PR in the first 16 weeks or SD for at least 16 weeks according to RECIST 1.1 by investigator assessment
Time to Response according to RECIST 1.1 by investigator assessment | Every 8 weeks (first 48 weeks) and then every 12 weeks from start of treatment until the earlier of progression, death or end of study (for max 42 months)
  Time from the start of study treatment until the date of first documented response (which is subsequently confirmed)
Best percentage change in tumour size according to RECIST 1.1 by investigator assessment | Every 8 weeks (first 48 weeks) and then every 12 weeks from start of treatment until the earlier of progression, death, start of subsequent anti-cancer therapy or end of study (for max 42 months)
  Best percentage change from baseline in sum of the diameters of target lesions
Overall Survival at 18 months | From start of treatment until the earlier of death or end of study (for max of 42 months). Each subject is followed for a minimum of 18 months and the landmark OS rate at 18 months will be estimated using a Kaplan-Meier analysis
  The survival rate of subjects at 18 months from start of treatment
Maximum concentration (Cmax) of AZD8701 in plasma when administered as monotherapy and in combination with Durvalumab | Cycle 1: Day 1, 2, 3, 5, 8. Cycle 2: Day 1, 22, 23. Cycle 3 & 4: Day 1 and at 105 day follow up (up to 28 months)
  Maximum concentration (Cmax) of AZD8701 in plasma
Time to maximum concentration (tmax) of AZD8701 in plasma when administered as monotherapy and in combination with Durvalumab | Cycle 1: Day 1, 2, 3, 5, 8. Cycle 2: Day 1, 22, 23. Cycle 3 & 4: Day 1 and at 105 day follow up (up to 28 months)
  Time to maximum concentration (tmax) of AZD8701 in plasma
Exposure to AZD8701 through measurement of area under the curve (AUC) in plasma when administered as monotherapy and in combination with Durvalumab | Cycle 1: Day 1, 2, 3, 5, 8. Cycle 2: Day 1, 22, 23. Cycle 3 & 4: Day 1 and at 105 day follow up (up to 28 months)
  Exposure to AZD8701 through measurement of area under the curve (AUC) in plasma
Maximum concentration (Cmax) of AZD8701 in urine when administered as monotherapy and in combination with Durvalumab | Cycle 1: Day 1, 2. Cycle 2: Day 22, 23 (up to 2 months)
  Maximum concentration (Cmax) of AZD8701 in urine
Time to maximum concentration (tmax) of AZD8701 in urine when administered as monotherapy and in combination with Durvalumab | Cycle 1: Day 1, 2. Cycle 2: Day 22, 23 (up to 2 months)
  Time to maximum concentration (tmax) of AZD8701 in urine
Exposure to AZD8701 through measurement of area under the curve (AUC) in urine when administered as monotherapy and in combination with Durvalumab | Cycle 1: Day 1, 2. Cycle 2: Day 22, 23 (up to 2 months)
  Exposure to AZD8701 through measurement of area under the curve (AUC) in urine
Urine concentrations of AZD8701 to assess renal clearance when administered as monotherapy and in combination with Durvalumab | Cycle 1: Day 1, 2. Cycle 2: Day 22, 23 (up to 2 months)
  Urine samples will be collected to assess urine concentrations of AZD8701 at a series of timepoints to derive renal clearance
Maximum concentration (Cmax) of Durvalumab in serum when administered in combination with AZD8701 | Cycle 1, 2, 3, 4 on Day 1 and 105 follow up (up to 28 months)
  Maximum concentration (Cmax) of Durvalumab in serum
Minimum concentration (Cmin) of Durvalumab in serum when administered in combination with AZD8701 | Cycle 1, 2, 3, 4 on Day 1 and 105 follow up (up to 28 months)
  Minimum concentration (Cmin) of Durvalumab in serum
Change in FOXP3 mRNA expression | From day 1 to day 29
  Percentage change in FOXP3 mRNA expression from pre-treatment (baseline) to post treatment

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Huntersville, North Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Madison, Wisconsin
- Research Site, Toronto, Ontario, Canada
- France (2):
  - Research Site, Rennes
  - Research Site, Villejuif
- Spain (3):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Revenko A, Carnevalli LS, Sinclair C, Johnson B, Peter A, Taylor M, Hettrick L, Chapman M, Klein S, Solanki A, Gattis D, Watt A, Hughes AM, Magiera L, Kar G, Ireland L, Mele DA, Sah V, Singh M, Walton J, Mairesse M, King M, Edbrooke M, Lyne P, Barry ST, Fawell S, Goldberg FW, MacLeod AR. Direct targeting of FOXP3 in Tregs with AZD8701, a novel antisense oligonucleotide to relieve immunosuppression in cancer. J Immunother Cancer. 2022 Apr;10(4):e003892. doi: 10.1136/jitc-2021-003892. PMID 35387780
- See also: Related Info — http://BreastCancerStudyLocator.com